CLINICAL TRIAL: NCT01801384
Title: Phase 2 Study of the Efficacy of Voucher-Based Incentives to Treat Pregnant Smokers
Brief Title: Voucher Based Incentives to Treat Pregnant Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Stephen T. Higgins, PhD, Professor of Psychiatry and Psychology, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01DA014028 (NIH)
Record Dates: First submitted 2013-02-26; First posted 2013-02-28 (Estimated); Last update posted 2023-05-12 (Actual); Status verified 2013-03

CONDITIONS: Efficacy of Financial Incentives
Keywords: pregnancy; cigarette smoking; incentives; smoking cessation; birth outcomes
MeSH Terms: conditions — Cigarette Smoking; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Original contingent vouchers schedule (Experimental): Women will receive an abstinence-contingent voucher-based incentives intervention (Contingency Management) for smoking cessation and relapse prevention.
  Interventions: Behavioral: Voucher-based incentives
- Revised contingent vouchers schedule (Experimental): Women receive abstinence-contingent voucher-based incentives (Contingency Management) intervention designed to further increase cessation and relapse prevention rates.
  Interventions: Behavioral: Voucher-based incentives
- Non-contingent vouchers schedule (Sham Comparator): This serves as a control condition wherein women earn incentives independent of smoking status.
  Interventions: Behavioral: Voucher-based incentives

INTERVENTIONS:
Behavioral: Voucher-based incentives
  Other Names: Contingency Management

SUMMARY:
The major goal of this project is to examine the efficacy of a voucher-based incentive program for promoting smoking cessation (Study 1) and preventing relapse (Study 2) during pregnancy and postpartum. Identifying efficacious interventions to increase cessation rates and decrease relapse among those who are able to quit is important to improving U.S. public health.

DETAILED DESCRIPTION:
Maternal cigarette smoking is the leading preventable cause of poor pregnancy outcomes and pediatric morbidity and mortality in the U.S. Efficacious interventions have been developed for smoking cessation during pregnancy, but cessation rates are low, typically under 20%. Efficacious interventions to prevent postpartum relapse remain to be developed. This application seeks support for a Stage II behavioral therapies development project to continue examining interventions to increase smoking cessation above the low levels noted above and to decrease postpartum relapse.

With regard to cessation, we conducted studies during the prior funding period showing that voucher-based incentives delivered contingent on biochemically-verified abstinence promote smoking cessation in approximately 40% of women who were still smoking at their 1st prenatal visit compared to only 9% in a control condition. Comparable studies on decreasing postpartum relapse among women who were smokers upon learning of their pregnancy but quit by their 1st prenatal visit (spontaneous quitters) supported the efficacy of abstinence-contingent vouchers for preventing antepartum but not postpartum relapse. We also completed secondary studies on appropriate cutpoints for biochemically verifying smoking status in pregnant women, characterizing the quantitative relationship between smoking exposure and fetal growth, the time-course of depressive symptoms during pregnancy in smokers and abstainers, and the incidence and severity of nicotine withdrawal.

While the treatment effect on smoking cessation during pregnancy noted above is at least two-fold greater than usual outcomes, the majority of women, especially heavier smokers (> 10 cigs/day), failed to quit. In Study 1 of this application we propose to experimentally examine whether a revised voucher program designed to increase initial abstinence and encourage additional quit attempts among those who initially fail can promote cessation at the end-of-pregnancy assessment in the majority of women treated (> 60%). Considering that nobody has succeeded in decreasing postpartum relapse among spontaneous quitters, we are not surprised that our first effort was unsuccessful. In Study 2 of this application we propose to experimentally test whether a revised voucher-based incentive program designed to more effectively reinforce sustained abstinence will decrease postpartum relapse. We are also proposing to continue secondary studies on biochemical verification of smoking status, fetal growth, and predictors of postpartum relapse.

Overall, the proposed studies have the potential to contribute important new information on effective treatments for one of our nation's most daunting drug abuse problems.

ELIGIBILITY:
Inclusion Criteria: Only women will participate in the proposed study, because the overarching aim is to develop efficacious treatments for smoking cessation and relapse prevention during pregnancy and early postpartum. All participants will be currently pregnant and report being smokers at the time of conception. Those in Study 1 will report continuing to smoke upon entering prenatal care. Those in Study 2 will report having already quit smoking upon entering prenatal care. Women must reside in the county in which the clinic is located, plan to reside in this geographical area through 6 months postpartum, be < 25 weeks gestation, not be living in a group residence, English speaking, and not regularly receiving psychotropics other than antidepressants.

-

Exclusion Criteria: Women receiving opioid substitution therapy will be excluded. In Vermont, minorities comprise 4% of the general population. There will be no exclusion criteria concerning race or ethnicity. In our studies during the prior funding period, approximately 5% of participants were minorities. We anticipate a similar sample in the proposed studies. We shall do all that we can to assure that minorities are included in the research.

-

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 166 (Actual)
Dates: Start 2006-04 (Actual); Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Biochemical verification of smoking status. | 15 months

SECONDARY OUTCOMES:
birth outcomes | 9 months
  Assessing the impact of smoking cessation on birth outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen T Higgins, Ph.D., Principal Investigator — University of Vermont
Locations (1):
- Substance Abuse Treatment Center, University of Vermont; UHC, Burlington, Vermont, United States

REFERENCES:
- [Background] Solomon LJ, Higgins ST, Heil SH, Badger GJ, Mongeon JA, Bernstein IM. Psychological symptoms following smoking cessation in pregnant smokers. J Behav Med. 2006 Apr;29(2):151-60. doi: 10.1007/s10865-005-9041-4. Epub 2006 Mar 14. PMID 16534659
- [Background] Higgins ST, Heil SH, Badger GJ, Mongeon JA, Solomon LJ, McHale L, Bernstein IM. Biochemical verification of smoking status in pregnant and recently postpartum women. Exp Clin Psychopharmacol. 2007 Feb;15(1):58-66. doi: 10.1037/1064-1297.15.1.58. PMID 17295585
- [Background] Solomon LJ, Higgins ST, Heil SH, Badger GJ, Thomas CS, Bernstein IM. Predictors of postpartum relapse to smoking. Drug Alcohol Depend. 2007 Oct 8;90(2-3):224-7. doi: 10.1016/j.drugalcdep.2007.03.012. Epub 2007 May 1. PMID 17475418
- [Background] Yoon JH, Higgins ST, Heil SH, Sugarbaker RJ, Thomas CS, Badger GJ. Delay discounting predicts postpartum relapse to cigarette smoking among pregnant women. Exp Clin Psychopharmacol. 2007 Apr;15(2):176-86. doi: 10.1037/1064-1297.15.2.186. PMID 17469941
- [Background] Heil SH, Higgins ST, Bernstein IM, Solomon LJ, Rogers RE, Thomas CS, Badger GJ, Lynch ME. Effects of voucher-based incentives on abstinence from cigarette smoking and fetal growth among pregnant women. Addiction. 2008 Jun;103(6):1009-18. doi: 10.1111/j.1360-0443.2008.02237.x. PMID 18482424
- [Background] Higgins ST, Chilcoat HD. Women and smoking: an interdisciplinary examination of socioeconomic influences. Drug Alcohol Depend. 2009 Oct 1;104 Suppl 1(Suppl 1):S1-5. doi: 10.1016/j.drugalcdep.2009.06.006. Epub 2009 Jul 8. No abstract available. PMID 19586726
- [Background] Higgins ST, Heil SH, Badger GJ, Skelly JM, Solomon LJ, Bernstein IM. Educational disadvantage and cigarette smoking during pregnancy. Drug Alcohol Depend. 2009 Oct 1;104 Suppl 1(Suppl 1):S100-5. doi: 10.1016/j.drugalcdep.2009.03.013. Epub 2009 May 12. PMID 19442460
- [Background] Linares Scott TJ, Heil SH, Higgins ST, Badger GJ, Bernstein IM. Depressive symptoms predict smoking status among pregnant women. Addict Behav. 2009 Aug;34(8):705-8. doi: 10.1016/j.addbeh.2009.04.003. Epub 2009 Apr 19. PMID 19411145
- [Result] Heil SH, Higgins ST, Mongeon JA, Badger GJ, Bernstein IM. Characterizing nicotine withdrawal in pregnant cigarette smokers. Exp Clin Psychopharmacol. 2006 May;14(2):165-70. doi: 10.1037/1064-1297.14.2.165. PMID 16756420
- [Result] Higgins ST, Heil SH, Dumeer AM, Thomas CS, Solomon LJ, Bernstein IM. Smoking status in the initial weeks of quitting as a predictor of smoking-cessation outcomes in pregnant women. Drug Alcohol Depend. 2006 Nov 8;85(2):138-41. doi: 10.1016/j.drugalcdep.2006.04.005. Epub 2006 May 23. PMID 16720082
- [Result] Heil, S.H., Yoon, J.H. & Higgins, S.T., (2008). Pregnant and Postpartum Women. In S.T. Higgins, K. Silverman, & S.H. Heil (Eds.), Contingency management in substance abuse treatment (pp. 182-201). New York, NY: The Guilford Press.
- [Derived] Higgins ST, Washio Y, Lopez AA, Heil SH, Solomon LJ, Lynch ME, Hanson JD, Higgins TM, Skelly JM, Redner R, Bernstein IM. Examining two different schedules of financial incentives for smoking cessation among pregnant women. Prev Med. 2014 Nov;68:51-7. doi: 10.1016/j.ypmed.2014.03.024. Epub 2014 Apr 2. PMID 24704135